CLINICAL TRIAL: NCT01051648
Title: Triamcinolone Assisted Anterior Vitrectomy in Complicated Cataract Surgery and Anterior Segment Reconstruction
Brief Title: Triamcinolone Assisted Anterior Vitrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: AL-Nour Eye Hospital (Other); Kasr El Aini Hospital (Other)
Responsible Party: Dr.Mostafa A EL-Helw,assistant. professor of Ophthalmology Cairo university, Cairo university medical school. EL-Nour Eye hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Triam1
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2008-02

CONDITIONS: Vitrectomy; Cataract
Keywords: Triamcinolone acetenoide; anterior vitrectomy; presence of vitreous in the anterior chamber.; effect of triamcinolone injection on IOP,intraocular infection
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Triamcinolone acetenoide (Experimental): Intra ocular injection of triamcinolone acetonide to visualize vitreous strands in the anterior chamber of the eye in complicated cataract surgery
  Interventions: Drug: Intra ocular injection of triamcinolone acetonide

INTERVENTIONS:
Drug: Intra ocular injection of triamcinolone acetonide — In all patients triamcinolone acetonide was prepared by keeping the bottle vertical to allow sedimentation of crystals thus removing the vehicle. It was then injected into the anterior chamber (2 ml with concentration 20 mg/ml) just prior to anterior vitrectomy. The direction of the tip of the needle was kept away from the corneal endothelium to minimize endothelial toxicity. Triamcinolone was removed as quickly & completely as possible after finishing anterior vitrectomy
  Other Names: kena cort

SUMMARY:
Injecting Triamcinolone acetenoide for visualizing and removing vitreous from the anterior chamber.

DETAILED DESCRIPTION:
The research followed the tenets of the Declaration of Helsinki, ;informed consent were obtained from patients where all details of the procedure were explained with emphasis on the intended outcome. The research was approved by the institutional review board.

Ten eyes of 10 patients were divided into 2 groups. Group A included 6 eyes of 6 patients with accidental rupture of posterior capsule during cataract surgery (5 eyes underwent phacoemulsification technique and one underwent ECCE). Group B included four eyes of 4 patients undergoing anterior segment reconstruction (anterior vitrectomy, secondary IOL Implantation and iris repair by direct approximation using 10/0 prolene sutures). In group A the mean age was 68.1 ± 10.93 years (range 47 to 79 years), 3 were males and 3 were females. In group B the mean age was 14 ± 5.6 years (range 9 to 22 years), 3 were males and one female. Demographic data and pre-operative Information are presented in table 1 and 2.

In all patients triamcinolone acetonide was prepared by keeping the bottle vertical to allow sedimentation of crystals thus removing the vehicle. It was then injected into the anterior chamber (2 ml with concentration 20 mg/ml) just prior to anterior vitrectomy. The direction of the tip of the needle was kept away from the corneal endothelium to minimize endothelial toxicity. Triamcinolone was removed as quickly & completely as possible after finishing anterior vitrectomy.

Postoperative regimen included topical steroids and antibiotics for about 4-6 weeks. Topical anti-glaucoma drugs were used in cases of high postoperative IOP for few days until stabilization of IOP. Follow up period ranged from 2 months up to 27 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vitreous in the anterior chamber whether in

  * complicated cataract surgery
  * disorganized anterior segment structures

Exclusion Criteria:

* Glaucoma patients
* Intra ocular infections
* Bacterial or fungal

Ages: 47 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Proper visualization of vitreous strands in the anterior chamber of the eye | immediately

SECONDARY OUTCOMES:
intraocular pressure rise | 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A EL-Helw, M.D., Principal Investigator — Cairo unuversity & EL-Nour eye hospital; Ahmed M Emarah, M.D., Principal Investigator — Cairo university & EL-Nour eye hospital
Locations (2):
- Egypt (2):
  - El-Nour Eye hospital, Cairo
  - Kasr Al-Ainy Hospital Cairo university, Cairo